CLINICAL TRIAL: NCT00793390
Title: A Case-Control Study of Inflammatory Breast Cancer in North Africa
Brief Title: Case-Control Study of Inflammatory Breast Cancer in North Africa
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909033; 09-C-N033
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Diabetes
Keywords: Aggressive Breat Cancer
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — saliva, tumor tissue

GROUPS / COHORTS (3):
- inflammatory breast cancer cases: inflammatory breast cancer cases
- non-inflammotory breast cancer cases: non-inflammatory breast cancer cases
- visitor controls without cancer: visitor controls without breast cancer- those visiting cancer patients

SUMMARY:
Background:

* Inflammatory breast cancer (IBC) is a rare, poorly understood and particularly aggressive form of breast cancer.
* Three characteristics of IBC tumors their rapid progression, their extensive formation of new blood vessels, and the fact that these characteristics are present from the inception of the tumor make it an ideal model for studying factors associated with tumor aggressiveness.
* This study is a collaboration among several institutions in the United States and North Africa that have extensive epidemiological experience and experience with IBC.

Objectives:

- To understand what causes certain types of breast conditions, including IBC.

Eligibility:

- Women 18 years of age and older with IBC and non-IBC and healthy women volunteers are eligible. Women who have had a previous diagnosis of any kind of breast cancer are excluded.

Design:

* Participants complete a questionnaire providing information about their background, including medical and reproductive history, family health history and lifestyle habits and undergo the following additional procedures:
* Height, weight, hip and chest measurements.
* Saliva sample collection to measure biological factors that may be related to breast conditions.
* Breast examination and, if permission is given, photographs of affected breast.
* Analysis of biopsied tissue for genetic and biochemical factors.

DETAILED DESCRIPTION:
Inflammatory breast cancer (IBC) is a rare, poorly understood and particularly aggressive form of breast cancer characterized by diffuse erythema and edema/peau d orange of the breast. The proposed case-control study of risk factors for IBC will include approximately 400 IBC cases accrued over a two-year period in centers in four countries in North Africa (the major cancer center and selected private clinicians in Tunisia, the major cancer center in Egypt, 2 cancer centers in Algeria, and 2 cancer centers in Morocco). Two control groups will be included: 1) 400 non-IBC breast cancer cases and; 2) 400 visitor controls (excluding those with breast, ovarian, endometrial, and nasopharyngeal cancers) in the study hospitals. The study will involve the administration of a questionnaire, anthropometric measurements, and saliva collection for all study subjects. In addition, digital photographs of the breasts will be collected for IBC cases, and a clinical examination form and paraffin-embedded tumor tissue will be collected for IBC cases and non-IOBC breast cancer controls. The study will be conducted as a consortium, with form development and translation coordinated at the National Cancer Institute (USA). A review of study procedures will be done after the first three months of data collection. The National Cancer Institute (NCI)-Division of Cancer Epidemiology and Genetics (DCEG), NCI-Office of International Affairs (OIA), University of Michigan, and International Breast Cancer Research Foundation (IBCRF) will provide funding for the project.

ELIGIBILITY:
* The case-control study will be restricted to women at least 18 years of age. IBC cases will be defined as having any clinical signs of redness, and either edema or peau d' orange characteristic of IBC or evidence of tumor emboli in the dermal lymphatics (at the center in Rabat).

Cases with extensive ulceration of the breast or with breast carcinoma 'en cuirasse' will be excluded from the study, even if erythema is present.

Women with a previous diagnosis of breast cancer will be excluded.

All cancers will be pathologically confirmed with evidence of tumor in either the breast parenchyma or dermal lymphatics based on the diagnostic biopsy.

Cases newly diagnosed and/or treated at study hospitals will be included.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at study hospitals and visitors to study hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 815 (Actual)
Dates: Start 2008-11-17 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
breast cancer | retrospective
  a rare type of breast cancer assessed clinically by study clinicians.

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Benson, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (6):
- Egypt (3):
  - National Cancer Institute-Cairo, Cairo
  - Gharbia Cancer Society, Gharbia
  - Tanta Cancer Center, Tanta
- Morocco (2):
  - Ibn Rochd Oncology Center, Casablanca
  - University Hospital Center Mohammed VI, Marrakesh
- Institut Salah Azaiz, Tunis, Tunisia